

# STUDY PROTOCOL

# **Study information**

| Title | Safety Profile of BNT162b2 mRNA SARS-Cov-2<br>Vaccine in Indonesia: A National Passive<br>Surveillance. |
|---|---|
| Protocol number | C4591050 |
| Protocol version identifier | Version 2.0 |
| Date | 26 April 2023 |
| Active substance | ATC code: J07BX03 Tozinameran - Nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2 |
| Medicinal product | BNT162b2 mRNA Vaccine |
| Research question and objectives | The objective of the study is to characterize descriptively the BNT162b2 vaccination experience among the Indonesian population, by analyzing structured data within Indonesia Vaccine Safety Databaseas requested by Indonesia Food and Drug Monitoring Agency (BPOM). |
| | Specific data elements include: |
| | A. Primary outcome measure : |
| | A1. SAE (Serious Adverse Event): SAE after primary dose and/or booster dose |
| | A2. Total AE reported after primary dose and/or booster dose |
| | B. Secondary outcome measure: |
| | B1. SAE onset : ≤30 mins or > 30 mins |

| | B2. Causality of SAE: coincidence, ISRR (Immunization Stress Related Response), vaccine reaction, unclassifiable, or indeterminate |
|---|---|
| | B3. Type of AE: |
| | B3.1. Serious and Non-serious |
| | B3.2. Solicited and unsolicited |
| | B4. Solicited AEs: |
| | B4.1 Local reactions : pain, swelling, redness, thickness. |
| | B4.2. Systemic reactions: fever, myalgia, malaise |
| | B5. Unsolicited AEs: |
| | B5.1. Local reactions: abscess, bleeding, etc. |
| | B5.2. Systemic reactions: headache, nausea, arthralgia, etc. |
| Author | PPD MD |
| Author | Pfizer MD |
| | PPD |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# 1. TABLE OF CONTENTS

| 1. TABLE OF CONTENTS | 3 |
|---|---|
| 2. LIST OF ABBREVIATIONS | 5 |
| 3. RESPONSIBLE PARTIES | 7 |
| 4. ABSTRACT | 8 |
| 5. AMENDMENTS AND UPDATES | 8 |
| 6. MILESTONES | 9 |
| 7. RATIONALE AND BACKGROUND | 9 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 10 |
| 9. RESEARCH METHODS | 10 |
| 9.1. Study design | 10 |
| 9.2. Setting. | 11 |
| 9.2.1. Inclusion criteria | 12 |
| 9.2.2. Exclusion criteria | 12 |
| 9.3. Variables | 12 |
| 9.4. Data sources | 13 |
| 9.5. Study size | 13 |
| 9.6. Data management | 14 |
| 9.7. Data analysis | 14 |
| 9.8. Quality control | 14 |
| 9.9. Limitations of the research methods | 14 |
| 9.10. Other aspects. | 14 |
| 10. PROTECTION OF HUMAN SUBJECTS | 15 |
| 10.1. Patient information | 15 |
| 10.2. Patient consent | 15 |
| 10.3. Patient withdrawal | 15 |
| 10.4. Institutional review board (IRB)/Independent ethics committee (IEC) | 15 |
| 10.5. Ethical conduct of the study | 15 |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 16 |
| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS PFIZER CONFIDENTIAL | 17 |

# BNT162b2 mRNA Vaccine C4591050 NON-INTERVENTIONAL STUDY PROTOCOL Version 2.0, Amendment 1,26 April 2023

| 13. REFERENCES | 17 |
|---------------------|----|
| 14. LIST OF TABLES | 18 |
| 15. LIST OF FIGURES | 18 |

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | Adverse event |
| BPOM | Indonesia Food and Drug Monitoring Agency |
| CIOMS | Council for International Organizations of Medical Sciences |
| COVID-19 | Coronavirus Disease 19 |
| EU | European Union |
| EUA | Emergency Use Authorization |
| FDA | Food and Drug Administration |
| GPP | Good Pharmacoepidemiology Practices |
| IBM-SPSS | Intelligence Based Manufacturing – Statistical Package of Social Science |
| IRB | Institutional Review Board |
| ISRR | Immunization Stress Related Response |
| IQR | Interquartiles Ranges |
| modRNA | Modified Ribonucleocid Acid |
| МоН | Ministry of Health |
| mRNA | Messenger Ribonucleic Acid |
| NCAEFI | National Committee of Adverse Event Following Immunization |
| NI | Non Interventional |
| SAE | Serious Adverse Events |

| SAP | Statistical Analysis Plan |
|------------|-------------------------------------------------|
| SARS-CoV-2 | Severe Acute Respiratory Syndrome Coronavirus 2 |
| WHO | World Health Organization |

# 3. RESPONSIBLE PARTIES

# **Principal Investigator(s) of the Protocol**

| Name, degree(s) | Job Title | Affiliation | Address |
|---|---|---|---|
| Dr. PPD | PPD | Pfizer | PPD |
| Dr. PPD | PPD | Pfizer | PPD |
| Dr. PPD | PPD | Pfizer | PPD |
| Dr. <b>PPD</b> PPD MSc-PH | PPD | NC AEFI (National<br>Committee of AE<br>Following<br>Immunizattion) | PPD |

# 4. ABSTRACT

None

# 5. AMENDMENTS AND UPDATES

| Amendment<br>number | Date | Protocol<br>section(s)<br>changed | Summary of amendment(s) | Reason |
|---|---|---|---|---|
| 1<br>administrative | 26 Apr<br>2023 | Section 6<br>MILESTONE<br>S | Modified Milestone | NA |
| | | Section 9<br>RESEARCH<br>METHODS | Deletion of text of SAP: Detailed<br>methodology for summary and<br>statistical analyses of data collected<br>in this study will be documented in a<br>statistical analysis plan (SAP),etc | Align with study team's decision. |

#### 6. MILESTONES

| Milestone | Planned date |
|--------------------------|---------------|
| Start of data collection | 16 March 2023 |
| End of data collection | 28 March 2023 |
| Final study report | 19 June 2023 |

#### 7. RATIONALE AND BACKGROUND

BPOM (Indonesia National Regulatory Authority) has issued an Emergency Use Authorization (EUA) to permit the emergency use of Comirnaty 30 mg/dose for primary and 15 mg/dose for booster concentrate for dispersion for injection. Comirnaty is indicated for active immunization to prevent COVID-19 caused by SARS-CoV-2 virus, in individuals 12 years of age and older in Indonesia. For detailed information please refer to the BPOM (Indonesia National Regulatory Authority) approved Fact Sheet For Health Care Providers EUA Of Comirnaty.

The safety of the primary series Pfizer-BioNTech COVID-19 Vaccine was evaluated in participants 6 months of age and older in 3 clinical studies conducted in the United States(US), Europe, Turkey, South Africa, and South America. Study BNT162-01 (Study 1) was a Phase 1/2, second-part, doseescalation trial that enrolled 60 participants, 18 through 55 years of age. Study C4591001 (Study 2) is a Phase 1/2/3, multicenter, multinational, randomized, saline placebo-controlled, observer-blind, dosefinding, vaccine candidate-selection (Phase 1) and efficacy (Phase 2/3) study that has enrolled approximately 46,000 participants, 12 years of age or older. Of these, approximately 43,448 participants [21,720 Pfizer-BioNTech COVID-19 Vaccine (30 mcg modRNA); 21,728 placebo] in Phase 2/3 are 16 years of age or older (including 138 and 145 participants 16 and 17 years of age in the vaccine and placebo groups, respectively) and 2,260 participants are 12 through 15 years of age (1,131 and 1,129 in the vaccine and placebo groups, respectively). Study C4591007 (Study 3) is a Phase 1/2/3 multicenter, randomized, dose-finding, open-label (Phase 1) and multinational, saline placebo-controlled, observer-blind, immunogenicity and efficacy (Phase 2/3) study that has enrolled 4,695 participants 5 through 11 years of age, of whom 3,109 participants received Pfizer-BioNTech COVID-19 Vaccine (10 mcg modRNA) and 1,538 participants received placebo in Phase 2/3. Study PFIZER CONFIDENTIAL

3 also enrolled 1,776 participants 6 through 23 months of age, of whom 1,178 participants were in the Pfizer-BioNTech COVID-19 Vaccine (3 mcg modRNA) group and 598 participants in the placebo group; and also enrolled 2,750 participants 2 through 4 years of age, of whom 1,835 participants were in the Pfizer-BioNTech COVID-19 Vaccine group and 915 participants in the placebo group in Phase 2/3. Results from these clinical studies have been published in peer-reviewed journals.

BPOM (Indonesia National Regulatory Authority) has requested to conduct an analysis of AEs reported in the Indonesia NC AEFI database following administration of BNT162b2 mRNA vaccine.

### 8. RESEARCH QUESTION AND OBJECTIVES

The objective of the study is to characterize descriptively the BNT162b2 vaccination safety experience among the Indonesian population, by analyzing structured data within Indonesia Vaccine Safety Website (Ministry of Health) as requested by BPOM (Indonesia National Regulatory Authority).

#### 9. RESEARCH METHODS

#### 9.1. Study design

This is a descriptive study for secondary data collection and analysis of structured data regarding AEs reported in Indonesia Vaccine Safety Website, following administration of primary and booster dose BNT162b2 mRNA vaccine. This study will not provide or make recommendations on any vaccine use.

- A. The AEs reported in Indonesia Vaccine Safety Database, following administration of BNT162b2 mRNA vaccine, are expected to be structured and anonymized/coded. Individual vaccine recipient identification information will not be collected in this study. The following data elements will be collected from the IndonesiaVaccine Safety Website for further analysis. Primary outcome measure:
  - A1. SAE (Serious Adverse Event): SAE after primary dose and/or booster dose
  - A2. Total AE reported after primary dose and/or booster dose
- B. Secondary outcome measure:
  - B1. SAE onset :  $\leq 30$  mins or  $\geq 30$  mins
  - B2. Causality of SAE: coincidence, ISRR (Immunization Stress Related Response), vaccine reaction, unclassifiable, or indeterminate

- B3. Type of AE:
  - B3.1. Serious and Non-serious
  - B3.2. Solicited and unsolicited
- **B4.** Solicited AEs:
  - B4.1.. Local reactions: pain, swelling, redness, thickness.
  - B4.2. Systemic reactions: fever, myalgia, malaise
- B5. Unsolicited AEs:
  - B5.1. Local reactions: abscess, bleeding, etc.
  - B5.2. Systemic reactions: headache, nausea, arthralgia, etc.

Since the study doesn't involve primary data collection from any participants, there will be no requirement of individual consent/ assent.

# 9.2. Setting

The secondary data collection will be exclusively from the Indonesia Vaccine Safety Website as requested by BPOM (Indonesia National Regulatory Authority). After the study protocol is approved by BPOM (Indonesia National Regulatory Authority), structured data will be obtained retrospectively for all AEs reported following administration of the BNT162b2 mRNA vaccine, starting from the time of vaccine available in Indonesia. Structured anonymized data for events which includes the following information will be collected and used for analysis:

- A. Primary outcome measure:
  - A1. SAE (Serious Adverse Event): SAE after primary dose and/or booster dose
  - A2. Total AE reported after primary dose and/or booster dose
- B. Secondary outcome measure:
  - B1. SAE onset :  $\leq 30$  mins or  $\geq 30$  mins
  - B2. Causality of SAE: coincidence, ISRR (Immunization Stress Related Response), vaccine reaction, unclassifiable, or indeterminate
  - B3. Type of AE:
    - B3.1. Serious and Non-serious
    - B3.2. Solicited and unsolicited
  - **B4.** Solicited AEs:

- B4.1.. Local reactions: pain, swelling, redness, thickness.
- B4.2. Systemic reactions: fever, myalgia, malaise
- B5. Unsolicited AEs:
  - B5.1. Local reactions: abscess, bleeding, etc.
  - B5.2. Systemic reactions: headache, nausea, arthralgia, etc.

Events for which either of the above is missing will not be recorded for analysis.

# 9.2.1. Inclusion criteria

This study will include adverse events reported in Indonesia NC AEFI database for individuals 12 years of age and older

#### 9.2.2. Exclusion criteria

The incomplete data in the database will be excluded

#### 9.3. Variables

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| The type of vaccination with BNT162b2 mRNA vaccine following which SAE was reported | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was<br>reported after primary<br>series or booster<br>vaccination |
| Onset of SAE | Baseline characteristic | Indonesia Vaccine<br>Safety Website | Whether the serious<br>AE onset ≤ 30 mins or<br>> 30 mins |
| Causality | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the SAE was caused by the vaccine. Causality of the AE with BNT162b2 – classified as WHO criteria as coincidence, ISRR, vaccine reaction, unclassifiable, or indeterminate) |
| Type of AE | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was<br>Serious and Non-<br>serious or solicited<br>and unsolicited |

| Type of solicited reaction | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was local or systemic |
|---|---|---|---|
| Type of Solicited<br>Local reaction | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was<br>pain, swelling, redness<br>or thickness |
| Type of Solicited<br>Systemic reaction | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was<br>fever, myalgia,<br>malaise |
| Type of unsolicited reaction | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was local or systemic and the term reported |
| Type of unsolicited local reaction | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was abscess, bleeding, etc. |
| Type of unsolicited systemic reaction | Baseline characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was<br>headache, nausea,<br>athralgia, fatigue, etc |
| Seriousness | Baseline<br>characteristics | Indonesia Vaccine<br>Safety Website | Whether the AE was serious according to Indonesia MoH decree (require hospitalization, life-threatening, cause persistent or significant disability/incapacity, or suspected to cause death) or non-serious |

# 9.4. Data sources

In Indonesia Vaccine Safety Website for AEs reported following administration of BNT162b2 mRNA vaccine

# 9.5. Study size

This is a descriptive study without a statistical hypothesis and hence sample size calculation is not applicable. In this study all the AEs reported following administration of BNT162b2 mRNA vaccine

will be collected retrospectively from the onset of this vaccine administration in Indonesia till the time of approval of this study.

#### 9.6. Data management

Data will be obtained from the Indonesia Vaccine Safety Website for AEs reported following administration of BNT162b2 mRNA vaccine as per the variables listed in section 9.3. A data management plan will be created before data collection begins and will describe all functions, processes, and specifications for data collection and analysis.

### 9.7. Data analysis

Descriptive Summary statistics will be presented to describe characteristics of events reports. Categorical covariates such as gender will be described by frequency distributions while continuous covariates such as age expressed will be summarized by in terms of their means and standard deviations or medians and interquartile ranges (IQR) as appropriate.

In addition, incidence rates will be computed as the number of events divided by the total number of vaccines administered.

All analyses will be done by Microsoft Excel

#### 9.8. Quality control

Not applicable

#### 9.9. Limitations of the research methods

This is a retrospective, observational study for secondary data collection and analysis of structured data regarding AEs reported in Indonesia NC AEFI database, following administration of BNT162b2 mRNA vaccine. The data availability will be contingent on the data provision by Indonesia NC AEFI post study approval by BPOM (Indonesia National Regulatory Authority). Since the data will originate and be owned by the Indonesia NC AEFI database, data validation and external quality control measures will not be applicable as a part of this study.

# 9.10. Other aspects

Not applicable

#### 10. PROTECTION OF HUMAN SUBJECTS

#### 10.1. Patient information

This study involves data that exist in anonymized structured format and contain no patient personal information.

### 10.2. Patient consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

#### 10.3. Patient withdrawal

Not applicable

# 10.4. Institutional review board (IRB)/Independent ethics committee (IEC)

There must be prospective approval of the study protocol, protocol amendments, and other relevant documents (e.g., informed consent forms if applicable) from the relevant IRBs/IECs. All correspondence with the IRB/IEC must be retained. Copies of IRB/IEC approvals must be forwarded to Pfizer.

# 10.5. Ethical conduct of the study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in

- Guidelines for Good Pharmacoepidemiology Practices (GPP). Public Policy
   Committee, International Society of Pharmacoepidemiology. Pharmacoepidemiology
   and Drug Safety
  - 2015; 25:2-10. https://onlinelibrary.wiley.com/doi/full/10.1002/pds.3891
- Good Practices for Outcomes Research issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR).
   http://www.ispor.org/workpaper/practices\_index.asp
- Good practices for real-world data studies of treatment and/or comparative effectiveness:
  - Recommendations from the joint ISPOR-ISPE Special Task Force on real-world evidence in

health care decision making.

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5639372/

- International Ethical Guidelines for Epidemiological Studies issued by the Council for International Organizations of Medical Sciences (CIOMS).
   https://cioms.ch/shop/product/international-ethical-guidelines-for-epidemiologicalstudies/
- European Medicines Agency (EMA) European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) Guide on Methodological Standards in Pharmacoepidemiology.
  - http://www.encepp.eu/standards\_and\_guidances/methodologicalGuide.shtml

Food and Drug Administration (FDA) Guidance for Industry: Good

Pharmacovigilance

Practices and Pharmacoepidemiologic Assessment.

https://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/

ucm071696.pdf

- FDA Guidance for Industry and FDA Staff: Best Practices for Conducting and Reporting Pharmacoepidemiologic Safety Studies Using Electronic Healthcare Data. http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidance
   s/UCM243537.pdf
- FDA Guidance for Industry: Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims.
   http://www.fda.gov/downloads/Drugs/Guidances/UCM193282.pdf

## 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the PFIZER CONFIDENTIAL

minimum criteria for reporting an AE (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

In the event of any prohibition or restriction imposed (eg, clinical hold) by an applicable competent authority in any area of the world, or if the investigator is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

#### 13. REFERENCES

- .
- 1. US FDA. Fact sheet for healthcare providers administering vaccine (vaccination providers): Emergency use authorization (EUA) of the Pfizer-Biontech COVID-19 vaccine to prevent coronavirus Disease 2019 (COVID-19); June 2022. https://www.fda.gov/media/159312/download accessed on 5 August 2022
- 2. BPOM. Fact Sheet For Health Care Providers Emergency Use Authorization (EUA) Of Comirnaty; July 2022.
- 3. Thomas SJ et al.; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine through 6 Months. N Engl J Med. 2021 Nov 4;385(19):1761-1773. doi: 10.1056/NEJMoa2110345. Epub 2021 Sep 15.
- Thomas S.J., et al. (2021). "Safety and Efficacy of the BNT162b2 mRNACovid-19 Vaccine through 6 Months." N Engl J Med. 385(19):1761-1773.
   Frenck, R. W., Jr., et al. (2021). "Safety, Immunogenicity, and Efficacy of the BNT162b2 Covid-19 Vaccine in Adolescents." N Engl J Med. 385(3): 239-250.
   Walter, E. B., et al. (2021). (2022) "Evaluation of the BNT162b2 Covid-19 Vaccine in Children 5 to 11 Years of Age." N Engl J Med. 386(1):35-46.
- 5. Frenck RW Jr et al.; C4591001 Clinical Trial Group. Safety, Immunogenicity, and Efficacy of the BNT162b2 Covid-19 Vaccine in Adolescents. N Engl J Med. 2021 Jul 15;385(3):239-250. doi: 10.1056/NEJMoa2107456. Epub 2021 May 27.

- 6. Polack FP et al.; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10.
- 7. Mulligan MJ et al. Phase I/II study of COVID-19 RNA vaccine BNT162b1 in adults. Nature. 2020 Oct;586(7830):589-593. doi: 10.1038/s41586-020-2639-4. Epub 2020 Aug 12. Erratum in: Nature. 2021 Feb;590(7844):E26.

#### 14. LIST OF TABLES

None

15. LIST OF FIGURES

None